CLINICAL TRIAL: NCT03057769
Title: Effect of Papillary Epinephrine Spraying on Post-ERCP Pancreatitis in Patients Received Rectal Indomethacin: A Multi-center, Double-blind, Randomized Controlled Trial
Brief Title: Effect of Papillary Epinephrine Spraying on Post-ERCP Pancreatitis in Patients Received Rectal Indomethacin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated because of an interim analysis suggesting futility of papillary epinephrine spraying in PEP prevention.
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associate professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20162097-1
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Pancreatitis; Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP, post-ERCP pancreatitis, indomethacin, epinephrine
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PES group (Experimental): All patients in this group receive 20 ml of 0.02% epinephrine sprayed on the duodenal papilla, over a period of 10-15 seconds using sphincterotome, at the end of procedure, just before the withdrawal of endoscope.
  Interventions: Drug: Papillary epinephrine spraying; Drug: Indomethacin
- Control group (Placebo Comparator): All patients in this group receive 20 ml of saline sprayed on the duodenal papilla, over a period of 10-15 seconds using sphincterotome, at the end of procedure, just before the withdrawal of endoscope.
  Interventions: Drug: Papillary saline spraying; Drug: Indomethacin

INTERVENTIONS:
Drug: Papillary epinephrine spraying — All patients in this group receive 20 ml of 0.02% epinephrine sprayed on the duodenal papilla, over a period of 10-15 seconds using sphincterotome, at the end of procedure, just before the withdrawal of endoscope.
  Other Names: PES
  Arms: PES group
Drug: Papillary saline spraying — All patients in this group receive 20 ml of saline sprayed on the duodenal papilla, over a period of 10-15 seconds using sphincterotome, at the end of procedure, just before the withdrawal of endoscope.
  Other Names: Control
  Arms: Control group
Drug: Indomethacin — All patients without contraindications should be administrated with rectal indomethacin within 30 min before ERCP.

SUMMARY:
Acute pancreatitis is the most common and feared complication of ERCP, occurring after 1% to 30% of procedures. It accounts for substantial morbidity and represents a substantial cost to health-care systems. European Society of Gastrointestinal Endoscopy and Japanese Society of Hepato-Biliary-Pancreatic surgery guidelines and recently large-scale RCT recommended routine use of NSAIDs indomethacin rectally before ERCP. Nonsteroidal anti-inflammatory drugs (NSAIDs) have been shown to inhibit prostaglandin synthesis, phospholipase A2 activity, and neutrophil/endothelial cell attachment, which is believed to play a key role in the pathogenesis of acute pancreatitis.

Other possible mechanisms have been suggested in the occurrence of pancreatitis. Papillary edema caused by manipulations during cannulation or endoscopic treatment has received the most attention. The papillary edema may cause temporary outflow obstruction of pancreatic juice, and then increase ductal pressure, resulting in the occurrence of pancreatitis. Topical application of epinephrine on the papilla may reduce papillary edema by decreasing capillary permeability or by relaxing the sphincter of Oddi. A meta-analysis (including 2 existing RCTs and post-hoc analysis of our previous study) of papillary epinephrine spraying compared with saline spraying or no intervention indicates a potential relative risk reduction of PEP (RR 0.34, 95%CI 0.19-0.61). Papillary epinephrine spraying may be an inexpensive and convenient alternative for prevention of post-ERCP pancreatitis. A large pragmatic RCT to determine whether routine using papillary epinephrine spraying can reduce post-ERCP pancreatitis is needed.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old patients planned for ERCP.

Exclusion Criteria:

* contraindications to ERCP
* allergy to epinephrine or NSAIDs
* Not suitable for pre-ERCP indomethacin (received NSAIDs within 7 days before the procedure; gastrointestinal hemorrhage within 4 weeks; renal dysfunction [Cr >1.4mg/dl=120umol/l]; presence of coagulopathy before the procedure)
* previous biliary sphincterotomy without planned pancreatic duct manipulation
* ERCP for biliary stent removal or exchange without planned pancreatic duct manipulation
* acute pancreatitis within 3 days before the procedure
* unwilling or inability to provide consent
* pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Overall post-ERCP pancreatitis (PEP) | 30 days

SECONDARY OUTCOMES:
Moderate to severe PEP | 30 days
Clinical significant gastrointestinal bleeding | 30 days
Overall ERCP complications | 30 days

OTHER OUTCOMES:
Severity of PEP evaluated by updated Atlanta criteria | 30 days
ERCP-related perforation | 30 days
Biliary infection | 30 days
Length of post-procedure hospital stay | 30 days
Death | 30 days

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Department of Gastroenterology, Successful Hospital of Xiamen university, Xiamen, Fujian
  - Department of Gastroenterology, Zhongshan Hospital of Xiamen university, Xiamen, Fujian
  - Department of General Surgery, The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Endoscopy Center, Ankang Central Hospital, Ankang, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Department of Gastroenterology, No. 451 Hospital, Xi'an, Shaanxi
  - Department of Gastroenterology, The First Affiliated Hospital of the Medical College, Shihezi University, Shihezi, Xinjiang
  - Department of Gastroenterology, Urumqi General Hospital of Lanzhou Military Region, Ürümqi, Xinjiang
  - Department of Gastroenterology, Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Department of Hepatobiliary Surgery, General Hospital of Ningxia Medical University, Yinchuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc. 2004 Jun;59(7):845-64. doi: 10.1016/s0016-5107(04)00353-0. No abstract available. PMID 15173799
- [Background] Dumonceau JM, Andriulli A, Elmunzer BJ, Mariani A, Meister T, Deviere J, Marek T, Baron TH, Hassan C, Testoni PA, Kapral C; European Society of Gastrointestinal Endoscopy. Prophylaxis of post-ERCP pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - updated June 2014. Endoscopy. 2014 Sep;46(9):799-815. doi: 10.1055/s-0034-1377875. Epub 2014 Aug 22. PMID 25148137
- [Background] Yokoe M, Takada T, Mayumi T, Yoshida M, Isaji S, Wada K, Itoi T, Sata N, Gabata T, Igarashi H, Kataoka K, Hirota M, Kadoya M, Kitamura N, Kimura Y, Kiriyama S, Shirai K, Hattori T, Takeda K, Takeyama Y, Hirota M, Sekimoto M, Shikata S, Arata S, Hirata K. Japanese guidelines for the management of acute pancreatitis: Japanese Guidelines 2015. J Hepatobiliary Pancreat Sci. 2015 Jun;22(6):405-32. doi: 10.1002/jhbp.259. Epub 2015 May 13. PMID 25973947
- [Background] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971
- [Background] Ding X, Chen M, Huang S, Zhang S, Zou X. Nonsteroidal anti-inflammatory drugs for prevention of post-ERCP pancreatitis: a meta-analysis. Gastrointest Endosc. 2012 Dec;76(6):1152-9. doi: 10.1016/j.gie.2012.08.021. PMID 23164513
- [Background] Matsushita M, Takakuwa H, Shimeno N, Uchida K, Nishio A, Okazaki K. Epinephrine sprayed on the papilla for prevention of post-ERCP pancreatitis. J Gastroenterol. 2009;44(1):71-5. doi: 10.1007/s00535-008-2272-8. Epub 2009 Jan 22. PMID 19159075
- [Background] Tarnasky P, Cunningham J, Cotton P, Hoffman B, Palesch Y, Freeman J, Curry N, Hawes R. Pancreatic sphincter hypertension increases the risk of post-ERCP pancreatitis. Endoscopy. 1997 May;29(4):252-7. doi: 10.1055/s-2007-1004185. PMID 9255527
- [Background] Johnson GK, Geenen JE, Johanson JF, Sherman S, Hogan WJ, Cass O. Evaluation of post-ERCP pancreatitis: potential causes noted during controlled study of differing contrast media. Midwest Pancreaticobiliary Study Group. Gastrointest Endosc. 1997 Sep;46(3):217-22. doi: 10.1016/s0016-5107(97)70089-0. PMID 9378207
- [Background] Ohno T, Katori M, Nishiyama K, Saigenji K. Direct observation of microcirculation of the basal region of rat gastric mucosa. J Gastroenterol. 1995 Oct;30(5):557-64. doi: 10.1007/BF02367779. PMID 8574325
- [Background] Xu LH, Qian JB, Gu LG, Qiu JW, Ge ZM, Lu F, Wang YM, Li YM, Lu HS. Prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis by epinephrine sprayed on the papilla. J Gastroenterol Hepatol. 2011 Jul;26(7):1139-44. doi: 10.1111/j.1440-1746.2011.06718.x. PMID 21392105
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Derived] Luo H, Wang X, Zhang R, Liang S, Kang X, Zhang X, Lou Q, Xiong K, Yang J, Si L, Liu W, Liu Y, Zhou Y, Wang S, Yang M, Chen W, Han Y, Shang G, Yang X, He Y, Zou Q, Guo W, Dai Y, Zeng W, Zhu X, Gong R, Li X, Nie Z, Wang Q, Wang L, Pan Y, Guo X, Fan D. Rectal Indomethacin and Spraying of Duodenal Papilla With Epinephrine Increases Risk of Pancreatitis Following Endoscopic Retrograde Cholangiopancreatography. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1597-1606.e5. doi: 10.1016/j.cgh.2018.10.043. Epub 2018 Oct 31. PMID 30391434